CLINICAL TRIAL: NCT01783639
Title: The WISE Study is a Pivotal Study Evaluating the Safety and Performance of WIRION™ EPD in Patients Undergoing Carotid Artery Stenting
Brief Title: Safety and Performance Evaluation of WIRION™ EPD in Patients Undergoing Carotid Artery Stenting
Acronym: WISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gardia Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: WIRION™ Pivotal Study (WISE); WIRION Study Europe (WISE) (Other: Gardia Medical Ltd.)
Record Dates: First submitted 2013-01-13; First posted 2013-02-05 (Estimated); Results first posted 2015-07-22 (Estimated); Last update posted 2017-08-07 (Actual); Status verified 2017-06

CONDITIONS: Carotid Artery Diseases; Stroke
Keywords: Carotid; Carotid artery stenting; Stent; Embolic protection; Atherosclerotic Disease
MeSH Terms: conditions — Carotid Artery Diseases; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Experimental): Device: WIRION™ Embolic Protection System
  Interventions: Carotid Artery Stent
  Interventions: Procedure: Carotid Artery Stent

INTERVENTIONS:
Procedure: Carotid Artery Stent — Assessment of the study device (WIRION) during carotid artery stenting procedure in comparison to a performance of FDA approved filter type embolic protection devices

SUMMARY:
The purpose of this study is to compare the safety and performance of WIRION™ EPD in patients undergoing carotid artery stenting to a performance goal based on an analysis of the results of previous US IDE carotid stenting with embolic protection studies

DETAILED DESCRIPTION:
Patient registry procedures include:

* Clinical Events Committee (CEC); responsibility for validating all reported primary safety outcomes
* Data Safety Monitoring Board (DSMB); to review and evaluate safety data including serious adverse events
* 100% data monitoring; to compare data entered into the registry
* Source data verification; to assess the accuracy, completeness of registry data by comparing the data to external data sources (e.g., medical records, paper or electronic case report forms).
* Standard Operating Procedures; to address registry operations and analysis activities, such as patient recruitment, data collection, data management, data analysis and reporting for adverse events.
* Sample size assessment to specify the number of participants and follow up duration.
* Data Management Plan; to address situations where variables are reported as missing, unavailable, "non-reported," uninterpretable, or considered missing because of data inconsistency or out-of-range results
* Statistical analysis plan; describing the analytical principles and statistical techniques to be employed in order to address the primary and secondary objectives, as specified in the study protocol or plan.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* Anticipated patient life expectancy of at least 1 year
* Patient or authorized representative, signed a written Informed Consent form
* Patient is willing to comply with the protocol requirements
* Candidate for catheter-based therapy of a single stenosis located in the internal carotid artery (ICA) or the carotid bifurcation, suitable for treatment with a single FDA-approved stent with a carotid use indication
* Reference vessel diameter for intended filter location between 3.5mm and 6.0mm
* An adequate "landing zone" of at least 30mm
* Patients with severe symptomatic or asymptomatic carotid artery stenosis, to be ≥ 50% for symptomatic patients OR ≥ 80% for asymptomatic patients
* At least one high surgical risk criteria, either anatomical or co-morbid risk factors, as listed below:

Category I - Anatomical high risk factors

* Recurrent stenosis after endarterectomy
* Previous radical neck surgery or radiation therapy to the neck
* High cervical ICA lesions or CCA lesions at or above C2 or below the clavicle
* Spinal immobility of the neck
* Tracheostomy or tracheal stoma
* Any laryngeal nerve palsy and bilateral carotid artery stenosis

Category II - Co-morbid risk factors

* Contralateral carotid occlusion
* Unstable angina (Canadian Cardiovascular Society class III/IV)
* Congestive Heart Failure (New York Heart Association functional class III/IV) and/or known severe left ventricular dysfunction LVEF<30%
* Requires coronary artery bypass surgery, cardiac valve surgery, major vascular surgery, or abdominal aortic aneurysm repair 31-60 days post carotid stent procedure
* Recent MI (>72 hr and <4 weeks)
* Severe pulmonary disease with FEV1 of <30%
* CAD in ≥2 unrevascularized vessels with stenosis ≥70%
* Age ≥75 years
* Uncontrolled diabetes - Female patient with no child bearing potential or has negative pregnancy test within the previous 7 days and agrees to remain on birth control throughout the study

Exclusion Criteria:

* Total occlusion or near-occlusion of the target vessel
* Severe lesion calcification
* Presence of an alternate source of emboli
* Presence of a filling defect, or angiographically visible thrombus, at target site
* A greater than 50% CCA lesion proximal to the target or a distal (intracranial) lesion more severe than the target lesion
* Evolving, acute or recent stroke within the last 30 days
* Major stroke with a residual neurological deficit that would confound neurologic assessment
* Vertebrobasilar insufficiency symptoms only
* Major operation 30 days before or after the index procedure
* Ipsilateral intracranial stenosis that requires treatment
* Any pre-existing stent in ipsilateral carotid artery, or placement of a stent in contralateral carotid within 30 days of the index procedure
* History of intracranial hemorrhage within 12 months
* Any condition that precludes proper angiographic assessment or prevents femoral arterial access
* Uncontrolled hypertension
* Contraindication to heparin and bivalirudin, aspirin, thienopyridines
* Known sensitivity to radiographic contrast media which cannot be controlled with pre-medication
* History or current indication of bleeding diathesis or coagulopathy
* Chronic renal insufficiency
* Carotid artery dissection or aortic arch anatomical anomalies
* Dementia or a neurological illness
* Patient is enrolled in another drug or device study protocol that has not reached its primary endpoint
* Severe pulmonary hypertension
* Intra-cranial pathology (e.g., tumor, AVM. aneurysm, etc) that would make study participation inappropriate or confound neurologic assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-02; Primary Completion 2013-12 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dierk Scheinert, MD, Principal Investigator — Herzzentrum Leipzig GmbH and Park-Krankenhaus Leipzig; Horst Sievert, MD, Principal Investigator — Cardio Vascular Center Frankfurt; Stefan Rohde, MD, Principal Investigator — Radiologische Klinik, Klinikum Dortmund GmbH; Joachim Schofer, MD, Principal Investigator — Universitäres Herz- und Gefäßzentrum Hamburg; Harald Mudra, MD, Principal Investigator — Städtisches Klinikum München GmbH; Marc Bosiers, MD, Principal Investigator — AZ St-Blasius, Dendermonde; Thomas Zeller, MD, Principal Investigator — Universitaets Herzzentrum, Bad-Krozingen; Alberto Cremonesi, MD, Principal Investigator — Villa Maria Cecilia, Contignola; Bernhard Reimers, MD, Principal Investigator — Mirano Hospital; Henrik Schröder, MD, Principal Investigator — Ihre-Radiologen.de
Locations (10):
- AZ Sint Blasius Hospital, Department of Vascular Surgery, Dendermonde, Belgium
- Germany (7):
  - Universitaets Herzzentrum, Bad Krozingen
  - Ihre-Radiologen.de, Berlin
  - Klinikum Dortmund GmbH, Dortmund
  - CardioVascular Center Frankfurt, Frankfurt
  - Hamburg University Cardiovascular Center, Hamburg
  - Herzzentrum and Park-Krankenhaus, Leipzig
  - Städtisches Klinikum München GmbH Klinikum Neuperlach, Munich
- Italy (2):
  - Villa Maria Cecilia Hospital, Cotignola
  - Mirano Hospital, Mirano

REFERENCES:
- [Derived] Scheinert D, Reimers B, Cremonesi A, Schmidt A, Sievert H, Rohde S, Schofer J, Mudra HG, Bosiers M, Zeller T, Pacchioni A, Rosenschein U; WISE (Wirion Study Europe) Pivotal Trial Investigators. Independent Modular Filter for Embolic Protection in Carotid Stenting. Circ Cardiovasc Interv. 2017 Mar;10(3):e004244. doi: 10.1161/CIRCINTERVENTIONS.116.004244. PMID 28283511

RESULTS

PARTICIPANT FLOW:
Groups:
- WIRION: Device: WIRION™ Embolic Protection System
  Interventions: Carotid Artery Stent
  Carotid Artery Stent: Assessment of the study device (WIRION) during carotid artery stenting procedure in comparison to a performance of FDA approved filter type embolic protection devices
Period: Overall Study
Arm/Group | WIRION
Started | 120
Completed | 120
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: Device: WIRION™ Embolic Protection System
  Interventions: Carotid Artery Stent
  Carotid Artery Stent: Assessment of the study device (WIRION) during carotid artery stenting procedure in comparison to a performance of FDA approved filter type embolic protection devices
Arm/Group | Arm 1
Number analyzed (Participants) | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 107
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.9 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 87
Region of Enrollment [Number; unit: participants]
  Belgium | 11
  Italy | 40
  Germany | 69

OUTCOME MEASURES:

1. Primary Outcome: The Rate of Peri-procedural (Within 30 Days of Procedure) Death, Stroke, and Myocardial Infarction.
Description: Each participant will be followed for 30 days of procedure during which the number of major cardiac and cerebral adverse events (Stroke, Death and Myocardial Infraction) will be counted to evaluate the device safety.
Time Frame: Within 30 Days of procedure
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Arm 1
Number analyzed (Participants) | 120
participants | 4 [0.9 to 8.3]

2. Secondary Outcome: The Rate of Device Success
Description: Defined as a successful delivery, deployment and retrieval of WIRION™ without any complications
Time Frame: Participants will be followed for the duration of the procedure, an expected average of 35 minutes
Reporting Status: Not Posted

3. Secondary Outcome: The Rate of Clinical Success
Description: Defined as freedom from procedure related serious adverse events
Time Frame: Participants will be followed for the duration of the procedure, an expected average of 35 minutes
Reporting Status: Not Posted

4. Secondary Outcome: The Rate of Access Site Complications
Time Frame: Within 30 Days of procedure
Reporting Status: Not Posted

5. Secondary Outcome: Neurological Events Occurring Within 30 Days Post Procedure,Including Strokes and Transient Ischemic Attacks
Time Frame: Within 30 Days of procedure
Reporting Status: Not Posted

6. Secondary Outcome: Angiographic Success
Description: Successful completion of the protected stent procedure without angiographic complications
Time Frame: Participants will be followed for the duration of the procedure, an expected average of 35 minutes
Reporting Status: Not Posted

7. Secondary Outcome: Procedural Success
Description: Defined as both device and angiographic success
Time Frame: Participants will be followed for the duration of the procedure, an expected average of 35 minutes
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | WIRION
Serious Adverse Events (participants affected / at risk) | 18/120
Other Adverse Events (participants affected / at risk) | 0/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | WIRION (N=120)
Neurological/ Nervous system (Nervous system disorders) | 7 (7)
Cardiovascular (Cardiac disorders) | 4 (4)
Low hemoglobin level (Blood and lymphatic system disorders) | 2 (2)
Severe anemia related to gastrointestinal bleeding (Gastrointestinal disorders) | 1 (1)
Admission at hospital with pain in segment L5/S1, protrusion of intervertebral discs (General disorders) | 1 (1)
Incomplete occulomoric paresis because of hypotension (General disorders) | 1 (1)
Macular artery occlusion (General disorders) | 1 (1)
Hospitalization due to aphasia and worsening of general health (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less